CLINICAL TRIAL: NCT01522417
Title: A Randomized, Multicenter, Open-Label Study to Evaluate the Efficacy of Tirofiban Using a High-Dose Bolus Plus a Shortened Infusion Duration Versus Label-Dosing Eptifibatide in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Shortened Aggrastat® Versus Integrilin in Percutaneous Coronary Intervention
Acronym: SAVI-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicure (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medicure 11002
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Infarction; Acute Coronary Syndromes; Unstable Angina
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Angina, Unstable | interventions — Tirofiban; Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Short Tirofiban (Aggrastat) (Experimental): Tirofiban (Aggrastat) will be dosed as a 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion during a PCI plus 1 to 2 hours post-PCI.
  Patients will receive tirofiban (Aggrastat) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Interventions: Drug: Short Tirofiban
- Eptifibatide (Integrilin) (Active Comparator): Eptifibatide (Integrilin) will be dosed as a 180 mcg/kg bolus followed by a 2.0 mcg/kg/min infusion for 12 to 18 hours, with a second 180 mcg/kg bolus 10 min after the first.
  Patients will receive eptifibatide (Integrilin) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Interventions: Drug: Eptifibatide
- Long Tirofiban (Aggrastat) (Experimental): Tirofiban (Aggrastat) will be dosed as a 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion for 12 to 18 hours post PCI.
  Patients will receive tirofiban (Aggrastat) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Interventions: Drug: Long Tirofiban

INTERVENTIONS:
Drug: Short Tirofiban — 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion during a PCI plus 1 to 2 hours post-PCI.
  Other Names: Aggrastat
  Arms: Short Tirofiban (Aggrastat)
Drug: Eptifibatide — 180 mcg/kg bolus followed by a 2.0 mcg/kg/min infusion for 12 to 18 hours, with a second 180 mcg/kg bolus 10 min after the first.
  Other Names: Integrilin
  Arms: Eptifibatide (Integrilin)
Drug: Long Tirofiban — 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion for 12 to 18 hours post-PCI.
  Other Names: Aggrastat
  Arms: Long Tirofiban (Aggrastat)

SUMMARY:
The purpose this study is to assess whether a tirofiban regimen of a high-dose bolus plus a shortened infusion duration compared to label-dosing eptifibatide in patients undergoing percutaneous coronary intervention (PCI) is associated with a non-inferior composite rate of death, PCI-related myocardial infarction, urgent target vessel revascularization or in-hospital major bleeding within 48 hours following PCI or hospital discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Scheduled to undergo PCI with an FDA, approved or cleared device (stent or procedures such as balloon angioplasty, rotoblation, AngioSculpt, laser atherectomy,etc.) in one or more native coronary target lesions
* Written informed consent

Exclusion Criteria:

* Primary PCI for STEMI as index procedure
* Prior STEMI within 48 hours before randomization
* Prior PCI within 30 days before randomization
* Planned staged PCI within the subsequent 24 hours after index PCI
* Use of abciximab within 7 days before randomization
* Use of tirofiban or eptifibatide within 12 hours before randomization
* Use of low-molecular weight heparin within 12 hours before randomization
* Use of bivalirudin within 12 hours before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2012-04; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven V Manoukian, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - North Georgia Heart Center, Gainesville, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Archbold Medical Center, Thomasville, Georgia
  - Lenox Hill Hospital, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Centennial Heart, Nashville, Tennessee
  - Chippenham Hospital, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first patient enrolled: 12 June 2012 ; Last patient completed 8 August 2018
  The study enrolled both stable and UA/NSTEMI patients scheduled to undergo PCI in one or more native coronary target lesions.
Pre-assignment Details: Decision to proceed to PCI, access site for PCI (transradial or transfemoral) and intended oral P2Y12 antagonist agent used post-randomization were all pre-specified prior to randomization to treatment groups.
Groups:
- Short Tirofiban (Aggrastat): Tirofiban (Aggrastat) will be dosed as a 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion during a PCI plus 1 to 2 hours post-PCI.
  Patients will receive tirofiban (Aggrastat) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Short Tirofiban: 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion during a PCI plus 1 to 2 hours post-PCI.
- Eptifibatide (Integrilin): Eptifibatide (Integrilin) will be dosed as a 180 mcg/kg bolus followed by a 2.0 mcg/kg/min infusion for 12 to 18 hours, with a second 180 mcg/kg bolus 10 min after the first.
  Patients will receive eptifibatide (Integrilin) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Eptifibatide: 180 mcg/kg bolus followed by a 2.0 mcg/kg/min infusion for 12 to 18 hours, with a second 180 mcg/kg bolus 10 min after the first.
- Long Tirofiban (Aggrastat): Tirofiban (Aggrastat) will be dosed as a 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion for 12 to 18 hours post PCI.
  Patients will receive tirofiban (Aggrastat) on a background of dual oral anti-platelet agents and unfractionated heparin (50 U/kg and repeat dosing per protocol guidelines).
  Long Tirofiban: 25 mcg/kg i.v. bolus followed by a 0.15 mcg/kg/min i.v. infusion for 12 to 18 hours post-PCI.
Period: Overall Study
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Started | 209 | 202 | 124 (Randomization into the long tirofiban arm was initiated on 14 June 2013.)
Completed | 209 | 202 | 124 (Randomization into the long tirofiban arm was completed on 1 February 2018.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) - all randomized patients who underwent PCI and received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat) | Total
Number analyzed (Participants) | 209 | 202 | 124 | 535
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.7) | 63.7 (10.1) | 62.6 (10.9) | 63.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 61 | 40 | 158
  Male | 152 | 141 | 84 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 3 | 17
  Not Hispanic or Latino | 202 | 195 | 121 | 518
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 27 | 20 | 18 | 65
  White | 175 | 173 | 103 | 451
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 209 | 202 | 124 | 535

OUTCOME MEASURES:

1. Primary Outcome: The Composite Endpoint of Death, Periprocedural Myonecrosis (PPM), Urgent Target Vessel Revascularization (uTVR) or Major Bleeding
Description: The composite of death (any-cause), periprocedural myonecrosis (defined as ≥ 3 times the upper limit of normal troponin and at least 20% or greater than the baseline troponin value), urgent target revascularization (repeat PCI or any CABG procedure after the index PCI on a non-selective basis in the target vessel because of recurrent myocardial ischemia) or non-CABG related major bleeding as quantified according to REPLACE-2 bleeding criteria.
Time Frame: 48 hours or hospital discharge, whichever came first
Population: As per the protocol, a patient must have a pre-PCI troponin measurement and at least one troponin measurement within 48 hours following PCI or hospital discharge, whichever comes first, otherwise they were excluded from the primary composite endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Number analyzed (Participants) | 202 | 194 | 123
Participants | 69 | 60 | 48

2. Secondary Outcome: The Composite Endpoint of Death, Periprocedural Myonecrosis or Urgent Target Vessel Revascularization
Description: The composite of death (any-cause), periprocedural myonecrosis (defined as ≥ 3 times the upper limit of normal troponin and at least 20% or greater than the baseline troponin value), or urgent target revascularization (repeat PCI or any CABG procedure after the index PCI on a non-selective basis in the target vessel because of recurrent myocardial ischemia)
Time Frame: 48 hours or hospital discharge, whichever came first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Number analyzed (Participants) | 202 | 194 | 123
Participants | 69 | 60 | 45

3. Secondary Outcome: Individual Components of Death, Urgent Target Revascularization or Major Bleeding
Description: Individual components of death (any-cause), urgent target revascularization (repeat PCI or any CABG procedure after the index PCI on a non-selective basis in the target vessel because of recurrent myocardial ischemia) or non-CABG related major bleeding as quantified according to REPLACE-2 major bleeding criteria.
Time Frame: 48 hours or hospital discharge, whichever came first
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Number analyzed (Participants) | 209 | 202 | 124
Participants
  Death | 0 | 1 | 0
  uTVR | 1 | 0 | 1
  REPLACE-2 Major Bleeding | 0 | 1 | 4

4. Secondary Outcome: Individual Components of Periprocedural Myonecrosis
Description: Individual components of periprocedural myonecrosis (PPM) (defined as ≥ 3 times, ≥ 10 times, ≥ 20 times or ≥ 50 times the upper limit of normal troponin and at least 20% or greater than the baseline troponin value)
Time Frame: 48 hours or hospital discharge, whichever came first
Population: As per the protocol, a patient must have a pre-PCI troponin measurement and at least one troponin measurement within 48 hours following PCI or hospital discharge, whichever comes first, otherwise they were excluded from the individual PPM endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Number analyzed (Participants) | 202 | 194 | 123
Participants
  ≥ 3 times ULN | 69 | 60 | 45
  ≥ 10 times ULN | 36 | 35 | 28
  ≥ 20 times ULN | 19 | 27 | 21
  ≥ 50 times ULN | 11 | 19 | 9

5. Secondary Outcome: The Composite Endpoint of Death, Periprocedural Myonecrosis (PPM) (≥ 10x Troponin), Urgent Target Vessel Revascularization (uTVR) or Major Bleeding
Description: The composite of death (any-cause), periprocedural myonecrosis (defined as ≥ 10 times the upper limit of normal troponin and at least 20% or greater than the baseline troponin value), urgent target revascularization (repeat PCI or any CABG procedure after the index PCI on a non-selective basis in the target vessel because of recurrent myocardial ischemia) or non-CABG related major bleeding as quantified according to REPLACE-2 bleeding criteria.
Time Frame: 48 hours or hospital discharge, whichever came first
Measure: Count of Participants; unit: Participants
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
Number analyzed (Participants) | 202 | 194 | 123
Participants | 36 | 35 | 32

ADVERSE EVENTS:
Time Frame: 48 hours or hospital discharge, whichever came first
Description: The Investigator periodically assessed patients for the occurrence of adverse events. To avoid bias in eliciting adverse events, patients were asked the following non-leading question: "How are you feeling?" All adverse events (serious and non-serious) reported by the patient will be followed until the event has resolved or has stabilized.
Arm/Group | Short Tirofiban (Aggrastat) | Eptifibatide (Integrilin) | Long Tirofiban (Aggrastat)
All-Cause Mortality (participants affected / at risk) | 0/209 | 1/202 | 0/124
Serious Adverse Events (participants affected / at risk) | 8/209 | 11/202 | 7/124
Other Adverse Events (participants affected / at risk) | 45/209 | 55/202 | 50/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Tirofiban (Aggrastat) (N=209) | Eptifibatide (Integrilin) (N=202) | Long Tirofiban (Aggrastat) (N=124)
Angina Pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary Artery Dissection (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Post-Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel Perforation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis in Device (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Tirofiban (Aggrastat) (N=209) | Eptifibatide (Integrilin) (N=202) | Long Tirofiban (Aggrastat) (N=124)
Catheter Site Haematoma (General disorders) | 7 (7) | 8 (8) | 4 (4)
Application Site Haemorrhage (General disorders) | 1 (1) | 5 (5) | 2 (2)
Infusion Site Haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel Puncture Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Troponin Increased (Investigations) | 8 (8) | 6 (6) | 4 (4)
Haematocrit Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Troponin T Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Glucose Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult Blood Positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin I Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0)
Coronary Artery Dissection (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Graft Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mental Status Change Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vascular Dissection (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel Perforation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Neurological Decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis in Device (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Testicular Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Randomization into the long tirofiban arm was initiated after 159 patients were already enrolled into either the short tirofiban or long eptifibatide arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT01522417/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT01522417/SAP_001.pdf